CLINICAL TRIAL: NCT03451331
Title: Randomized Phase 2 Trial of Gemcitabine + Carboplatin + Nivolumab Versus Gemcitabine + Oxaliplatin + Nivolumab in Cisplatin-ineligible Patients With Metastatic Urothelial Cancer
Brief Title: Gemcitabine + Carboplatin + Nivolumab Versus Gemcitabine + Oxaliplatin + Nivolumab in Cisplatin-ineligible Patients With Metastatic Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Matthew Galsky (Other)
Collaborators: Bristol-Myers Squibb (Industry); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor-Investigator, Matthew Galsky, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU16-287
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Urothelial Cancer
Keywords: cisplatin-ineligible; gemcitabine; carboplatin; nivolumab; oxaliplatin
MeSH Terms: interventions — Nivolumab; Gemcitabine; Carboplatin; Oxaliplatin

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (Experimental): Gemcitabine plus carboplatin plus nivolumab
  Interventions: Drug: Nivolumab; Drug: Gemcitabine; Drug: Carboplatin
- Arm B (Experimental): Gemcitabine plus oxaliplatin plus nivolumab
  Interventions: Drug: Nivolumab; Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 360mg (and/or) Maintenance Single Agent Nivolumab 480mg (starting ~ 2-4 weeks after completing combination chemotherapy plus nivolumab)
  Other Names: OPDIVO®
Drug: Gemcitabine — 1000 mg/m^2
  Other Names: Gemzar
Drug: Carboplatin — AUC 4.5 (based on the Calvert formula)
  Other Names: Paraplatin®
  Arms: Arm A
Drug: Oxaliplatin — 130 mg/m^2
  Other Names: Eloxatin
  Arms: Arm B

SUMMARY:
This is a randomized phase 2 trial of gemcitabine + carboplatin + nivolumab or gemcitabine + oxaliplatin + nivolumab for the treatment of cisplatin-ineligible patients with metastatic urothelial cancer. Randomization will be stratified on the lymph node only (and/or unresectable primary) metastatic status.

DETAILED DESCRIPTION:
Patients will be randomized to Arm A: gemcitabine plus carboplatin plus nivolumab versus Arm B: gemcitabine plus oxaliplatin plus nivolumab. Randomization will be stratified on the metastasis status (lymph node only vs. the rest). Patients on both treatment arms will receive up to 6 cycles of combination therapy in the absence of prohibitive adverse effects or disease progression. Patients with at least stable disease at the completion of 6 cycles of treatment may continue "maintenance" single agent nivolumab for up to 12 cycles. Patients who require discontinuation of chemotherapy (i.e., gemcitabine plus carboplatin or gemcitabine plus oxaliplatin) prior to Cycle 6, but who have at least stable disease, may be considered for ongoing treatment with single-agent nivolumab on the "maintenance" phase after discussion with the sponsor-investigator.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all the following applicable inclusion criteria to participate in this study:

* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of = 2
* Able to comply with the study protocol, in the investigator's judgment.
* Histologically documented, locally advanced (T4b, any N; or any T, N 2-3) or metastatic urothelial carcinoma (mUC) (M1, Stage IV) (also termed TCC or UCC of the urinary tract; including renal pelvis, ureters, urinary bladder, and urethra) Patients with mixed histologies are required to have a dominant transitional cell pattern. Locally advanced bladder cancer must be inoperable on the basis of involvement of pelvic sidewall or adjacent viscera (clinical Stage T4b) or bulky nodal metastasis (N2-N3).
* Measurable disease, as defined by RECIST v1.1
* Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens (metastatic specimens preferable but if not available primary tumor specimens that are at least muscle-invasive are acceptable) in paraffin blocks (blocks preferred) or at least 15 unstained slides. If archival tissue is not available, subjects may be considered for enrollment on a case by case basis after discussion with the sponsor-investigator.
* No prior chemotherapy for inoperable locally advanced or mUC. For patients who received prior adjuvant/neoadjuvant chemotherapy or chemo-radiation for urothelial carcinoma, a treatment-free interval > 12 months between the last treatment administration and the date of recurrence is required in order to be considered treatment naive in the metastatic setting.
* Cisplatin-ineligible as defined by at least one of the following:

  * Calculated creatinine clearance ≥ 30 (Cockroft-Gault)
  * ECOG performance status of 2 or greater
  * CTCAE v4 Grade ≥ 2 audiometric hearing loss
* Demonstrate adequate organ function. All screening labs to be obtained within 28 days prior to registration:

  * Hematological:

    * Absolute Neutrophil Count (ANC) ≥ 1.5 x 10^9/L
    * Hemoglobin (Hgb) ≥ 9 g/dL
    * Platelets ≥ 100 x 10^9/L
  * Renal:

    • Calculated creatinine clearance ≥ 30 mL/min (Cockroft-Gault)
  * Hepatic:

    * Bilirubin ≤ 1.5 × upper limit of normal (ULN) (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
    * Aspartate aminotransferase (AST) ≤ 3 × ULN
    * Alanine aminotransferase (ALT) ≤ 3 × ULN
* Women of childbearing potential must have a negative serum or urine pregnancy.
* Women of childbearing potential (WOCBP) and male subjects must use appropriate method(s) of contraception as stated for the timeline below. Male subjects are not required to use contraception as outlined in protocol.

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

* Active infection requiring systemic therapy.
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Any serious or uncontrolled medical disorder that, in the opinion of the site investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured.
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
* Grade ≥ 2 neuropathy (NCI CTCAE version 4).
* Known positive result for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (RNA) or hepatitis C antibody (HCV antibody) indicating acute or chronic infection. Testing at screening is not required.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class III or greater), myocardial infarction within 3 months prior to randomization, unstable arrhythmias, or unstable angina.
* Known left ventricular ejection fraction (LVEF) < 40% Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF 40%-50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
* Solid organ or tissue transplant including stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Galsky, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai; Tisch Cancer Institute
Locations (6):
- United States (6):
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - John Theuer Cancer Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Icahn School of Medicine: Tisch Cancer Institute at Mount Sinai Medical Center, New York, New York
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Huntsman Cancer Institute University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galsky MD, Daneshmand S, Izadmehr S, Gonzalez-Kozlova E, Chan KG, Lewis S, Achkar BE, Dorff TB, Cetnar JP, Neil BO, D'Souza A, Mamtani R, Kyriakopoulos C, Jun T, Gogerly-Moragoda M, Brody R, Xie H, Nie K, Kelly G, Horowitz A, Kinoshita Y, Ellis E, Nose Y, Ioannou G, Cabal R, Del Valle DM, Haines GK, Wang L, Mouw KW, Samstein RM, Mehrazin R, Bhardwaj N, Yu M, Zhao Q, Kim-Schulze S, Sebra R, Zhu J, Gnjatic S, Sfakianos J, Pal SK. Gemcitabine and cisplatin plus nivolumab as organ-sparing treatment for muscle-invasive bladder cancer: a phase 2 trial. Nat Med. 2023 Nov;29(11):2825-2834. doi: 10.1038/s41591-023-02568-1. Epub 2023 Oct 2. PMID 37783966
- See also: Hoosier Cancer Research Network Website — http://www.hoosiercancer.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 25 | 24
Completed | 23 | 23
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Unable to start treatment. | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 72 [65 to 78] | 72 [67 to 78] | 72 [66 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 18 | 16 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 22 | 21 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 19 | 17 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46
Tobacco use history [Count of Participants; unit: Participants]
  Never | 6 | 10 | 16
  Current | 1 | 2 | 3
  Former | 16 | 11 | 27
Primary tumor site [Count of Participants; unit: Participants]
  Bladder | 17 | 18 | 35
  Urethra | 3 | 2 | 5
  Renal pelvis | 2 | 2 | 4
  Ureters | 1 | 1 | 2
ECOG performance status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction, 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work, 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours and 5=Dead.
  Participants
    ECOG = 0 | 8 | 7 | 15
    ECOG = 1 | 11 | 8 | 19
    ECOG = 2 | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  ORR is defined as the percentage of patients who achieve a response (confirmed PR or CR) according to RECIST 1.1.
Time Frame: Up to a maximum of 50 months
Population: Out of 23 subjects in Arm B, two subjects were not evaluable for best response.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 23 | 21
Percentage of participants | 69.6 [47 to 87] | 33.3 [15 to 57]

2. Secondary Outcome: Adverse Events
Description: The frequency and severity of grade 3+ treatment emergent adverse events are reported by CTCAEv4 term and grade.
Time Frame: AE had been recorded from time of signed informed consent until 30 days after discontinuation of study drug(s) or until a new anti-cancer treatment starts, whichever occurs first, up to a maximum of 19 months.
Measure: Number; unit: Number of Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 23 | 23
Number of Participants
  Anemia | 8 | 3
  Febrile neutropenia | 2 | 0
  Hepatitis viral | 1 | 0
  Kidney infection | 2 | 0
  Lung infection | 1 | 0
  Other infections and infestations | 1 | 0
  Skin infection | 1 | 2
  Urinary tract infection | 4 | 1
  Alanine aminotransferase increased | 1 | 1
  Alkaline phosphatase increased | 0 | 2
  Aspartate aminotransferase increased | 1 | 4
  Lipase increased | 3 | 7
  Lymphocyte count decreased | 3 | 1
  Neutrophil count decreased | 12 | 6
  Other investigations | 1 | 0
  Platelet count decreased | 1 | 5
  Serum amylase increased | 1 | 4
  White blood cell decreased | 4 | 2
  Hyperglycemia | 0 | 1
  Hyponatremia | 1 | 0
  Hypophosphatemia | 1 | 0
  Muscle weakness left-sided | 1 | 0
  Peripheral sensory neuropathy | 1 | 0
  Atrial fibrillation | 1 | 0
  Bladder spasm | 1 | 0
  Dyspnea | 2 | 1
  Other respiratory, thoracic and mediastinal disorders | 1 | 2
  Other skin and subcutaneous tissue disorders | 2 | 0
  Rash maculo-papular | 2 | 0
  Other surgical and medical procedures | 0 | 1
  Hypertension | 1 | 2
  Hypotension | 1 | 0
  Thromboembolic event | 2 | 1
  Hearing impaired | 1 | 1
  Diarrhea | 0 | 1
  Nausea | 0 | 1
  Other gastrointestinal disorders | 0 | 1
  Pancreatitis | 1 | 0
  Upper gastrointestinal hemorrhage | 1 | 0
  Vomiting | 0 | 1
  Fatigue | 1 | 0
  Pain | 2 | 1

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the period measured from the date that evaluation criteria were met for CR or PR (whichever status was recorded first) until the date that recurrence or PD was objectively documented.
Time Frame: Up to a maximum of 50 months
Population: Out of 23 subjects in Arm B, two subjects were not evaluable for efficacy analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 23 | 21
Months | 8.64 [4.37 to 19.29] | 6.51 [1.2 to NA] — Not enough participants achieved response to calculate upper 95% confidence interval.

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD. PFS is defined as time from registration until disease progression met by RECIST 1.1 or death from any cause.
Time Frame: Up to maximum of 50 months
Population: Out of 23 subjects in Arm B, two subjects were not evaluable for efficacy analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 23 | 21
Months | 9.4 [5.62 to 12.88] | 8.57 [2.56 to 10.38]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization until death or date of last contact.
Time Frame: Up to a maximum of 53 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 23 | 23
Months | 24.74 [17.45 to NA] — Not enough events occur to calculate the upper 95% Confidence Interval. | 16.43 [7.66 to 28.68]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to a maximum of 53 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored up to 19 months.
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 12/23 | 16/23
Serious Adverse Events (participants affected / at risk) | 15/23 | 17/23
Other Adverse Events (participants affected / at risk) | 22/23 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=23) | Arm B (N=23)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (2) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (2) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
HEPATITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 1 (1) | 0 (0)
KIDNEY INFECTION (Infections and infestations) | 1 (1) | 0 (0)
MUSCLE WEAKNESS LEFT-SIDED (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
SKIN INFECTION (Infections and infestations) | 1 (1) | 2 (2)
STROKE (Nervous system disorders) | 1 (1) | 0 (0)
THROMBOEMBOLIC EVENT (Vascular disorders) | 2 (3) | 1 (1)
UPPER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 5 (8) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1)
BLADDER PERFORATION (Renal and urinary disorders) | 0 (0) | 1 (1)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CPK INCREASED (Investigations) | 0 (0) | 2 (3)
DIARRHEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
FEVER (General disorders) | 0 (0) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
INTRACRANIAL HEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1)
LIPASE INCREASED (Investigations) | 0 (0) | 1 (1)
PAIN (General disorders) | 0 (0) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 3 (4)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=23) | Arm B (N=23)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (4) | 4 (5)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 3 (3) | 1 (1)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (1) | 0 (0)
AGITATION (Psychiatric disorders) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 9 (15) | 14 (28)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 6 (8) | 7 (15)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
ANEMIA (Blood and lymphatic system disorders) | 19 (65) | 13 (27)
ANOREXIA (Metabolism and nutrition disorders) | 6 (6) | 13 (19)
ANXIETY (Psychiatric disorders) | 1 (1) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 7 (13) | 15 (46)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 (8) | 3 (3)
BLADDER INFECTION (Infections and infestations) | 1 (1) | 0 (0)
BLADDER SPASM (Renal and urinary disorders) | 1 (1) | 1 (1)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 3 (5) | 1 (2)
BLOOD BILIRUBIN INCREASED (Investigations) | 3 (3) | 1 (2)
BLURRED VISION (Eye disorders) | 1 (1) | 1 (1)
CARDIAC TROPONIN I INCREASED (Investigations) | 1 (1) | 0 (0)
CHILLS (General disorders) | 1 (1) | 2 (2)
CHOLESTEROL HIGH (Investigations) | 1 (1) | 0 (0)
CONDUCTION DISORDER (Cardiac disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 7 (10) | 9 (9)
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 4 (5)
CREATININE INCREASED (Investigations) | 7 (17) | 12 (19)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 1 (3)
DEPRESSION (Psychiatric disorders) | 1 (2) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 7 (9) | 14 (23)
DIZZINESS (Nervous system disorders) | 2 (2) | 3 (3)
DRY MOUTH (Gastrointestinal disorders) | 4 (4) | 2 (2)
DRY SKIN (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
DYSGEUSIA (Nervous system disorders) | 5 (6) | 3 (4)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 3 (4)
EAR PAIN (Ear and labyrinth disorders) | 1 (2) | 0 (0)
EDEMA FACE (General disorders) | 1 (1) | 0 (0)
EDEMA LIMBS (General disorders) | 3 (3) | 3 (3)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (6)
EYE DISORDERS - OTHER, SPECIFY (Eye disorders) | 1 (1) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
FATIGUE (General disorders) | 13 (23) | 14 (21)
FECAL INCONTINENCE (Gastrointestinal disorders) | 1 (1) | 1 (1)
FEVER (General disorders) | 8 (9) | 5 (6)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 0 (0)
FLU LIKE SYMPTOMS (General disorders) | 1 (1) | 0 (0)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 4 (4) | 1 (1)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 3 (3) | 4 (4)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 3 (3) | 3 (3)
HEADACHE (Nervous system disorders) | 2 (2) | 2 (2)
HEARING IMPAIRED (Ear and labyrinth disorders) | 1 (1) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 2 (3) | 3 (3)
HEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 1 (1)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 3 (4) | 9 (29)
HYPERKALEMIA (Metabolism and nutrition disorders) | 4 (10) | 4 (4)
HYPERSOMNIA (Nervous system disorders) | 1 (2) | 0 (0)
HYPERTENSION (Vascular disorders) | 3 (5) | 6 (8)
HYPERTHYROIDISM (Endocrine disorders) | 3 (3) | 2 (2)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 9 (16) | 10 (18)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (4) | 3 (9)
HYPONATREMIA (Metabolism and nutrition disorders) | 6 (9) | 4 (7)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 1 (2) | 2 (3)
HYPOTENSION (Vascular disorders) | 1 (2) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 3 (3) | 4 (4)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 1 (3) | 1 (1)
INJECTION SITE REACTION (General disorders) | 1 (1) | 1 (1)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
INSOMNIA (Psychiatric disorders) | 1 (1) | 5 (7)
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 2 (3) | 1 (1)
KIDNEY INFECTION (Infections and infestations) | 1 (1) | 0 (0)
LIPASE INCREASED (Investigations) | 4 (14) | 11 (28)
LOCALIZED EDEMA (General disorders) | 2 (3) | 0 (0)
LUNG INFECTION (Infections and infestations) | 2 (3) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 8 (28) | 8 (16)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 2 (2) | 2 (2)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 10 (11) | 14 (21)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (3)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 1 (1) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 17 (48) | 10 (39)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0)
PAIN (General disorders) | 9 (12) | 8 (11)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 (8) | 4 (6)
PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0)
PAPULOPUSTULAR RASH (Infections and infestations) | 1 (1) | 1 (1)
PERIORBITAL EDEMA (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 2 (2) | 2 (2)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (2) | 11 (18)
PHOTOSENSITIVITY (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 12 (38) | 17 (62)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 5 (7) | 5 (6)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 10 (16) | 4 (4)
RECTAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 2 (3) | 2 (2)
REPRODUCTIVE SYSTEM AND BREAST DISORDERS - OTHER, SPECIFY (Reproductive system and breast disorders) | 1 (1) | 0 (0)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
SERUM AMYLASE INCREASED (Investigations) | 6 (17) | 11 (33)
SINUS PAIN (Nervous system disorders) | 1 (2) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 7 (15) | 3 (4)
SKIN INFECTION (Infections and infestations) | 2 (4) | 3 (5)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
SURGICAL AND MEDICAL PROCEDURES - OTHER, SPECIFY (Surgical and medical procedures) | 3 (7) | 3 (4)
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 1 (2) | 0 (0)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 3 (3) | 0 (0)
URINARY FREQUENCY (Renal and urinary disorders) | 2 (3) | 4 (4)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (2) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (4) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 5 (6) | 4 (6)
URINARY TRACT PAIN (Renal and urinary disorders) | 2 (2) | 2 (2)
URINARY URGENCY (Renal and urinary disorders) | 1 (2) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (2) | 0 (0)
WATERING EYES (Eye disorders) | 1 (2) | 0 (0)
WEIGHT LOSS (Investigations) | 2 (2) | 6 (7)
WHITE BLOOD CELL DECREASED (Investigations) | 13 (46) | 10 (33)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 1 (1)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BLOATING (Gastrointestinal disorders) | 0 (0) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BRUISING (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 0 (0) | 1 (1)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 0 (0) | 1 (1)
CONFUSION (Psychiatric disorders) | 0 (0) | 1 (1)
CPK INCREASED (Investigations) | 0 (0) | 2 (4)
DRY EYE (Eye disorders) | 0 (0) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSESTHESIA (Nervous system disorders) | 0 (0) | 1 (3)
EYE PAIN (Eye disorders) | 0 (0) | 1 (1)
FLUSHING (Vascular disorders) | 0 (0) | 1 (1)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (7)
GLAUCOMA (Eye disorders) | 0 (0) | 1 (1)
GLUCOSE INTOLERANCE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HEMOGLOBIN INCREASED (Investigations) | 0 (0) | 1 (1)
HEPATOBILIARY DISORDERS - OTHER, SPECIFY (Hepatobiliary disorders) | 0 (0) | 2 (3)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HOT FLASHES (Vascular disorders) | 0 (0) | 2 (2)
HYPERNATREMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
HYPOKALEMIA (Metabolism and nutrition disorders) | 0 (0) | 4 (7)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
INR INCREASED (Investigations) | 0 (0) | 1 (1)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 1 (1)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
PARESTHESIA (Nervous system disorders) | 0 (0) | 2 (2)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 2 (2)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 2 (3)
SINUS DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 2 (2)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SUPERFICIAL THROMBOPHLEBITIS (Vascular disorders) | 0 (0) | 3 (3)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 2 (2)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 1 (1)
TREMOR (Nervous system disorders) | 0 (0) | 1 (1)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 2 (2)
VAGINAL FISTULA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VAGINAL HEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/31/NCT03451331/Prot_SAP_000.pdf